CLINICAL TRIAL: NCT02683200
Title: Stereotactic Body Radiotherapy for Liver Metastases and Hepatocellular Carcinoma Utilizing an MRI-Guided Tri-60Co Teletherapy System
Brief Title: MRI-Guided Stereotactic Body Radiation Therapy in Treating Patients With Liver Metastases or Liver Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-000362; NCI-2015-01665 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2015-10-09; First posted 2016-02-17 (Estimated); Last update posted 2023-02-21 (Actual); Status verified 2022-03

CONDITIONS: Adult Hepatocellular Carcinoma; Metastatic Malignant Neoplasm in the Liver
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes

ARMS (1):
- Treatment (MRI-guided Tri-60Co teletherapy SBRT) (Experimental): Patients undergo MRI-guided Tri-60Co teletherapy SBRT 3-5 fractions over 1-2 weeks.
  Interventions: Radiation: Image-Guided Adaptive Radiation Therapy; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Radiation: Image-Guided Adaptive Radiation Therapy — Undergo MRI-guided Tri-60Co teletherapy SBRT
  Other Names: IGART
Radiation: Stereotactic Body Radiation Therapy — Undergo MRI-guided Tri-60Co teletherapy SBRT
  Other Names: SBRT

SUMMARY:
This pilot clinical trial studies magnetic resonance imaging (MRI)-guided stereotactic body radiation therapy (SBRT) in treating patients with liver metastases or liver cancer. SBRT is a specialized radiation therapy that delivers a single, high dose of radiation directly to the tumor and may kill more tumor cells and cause less damage to normal tissue. Combining MRI with SBRT may help doctors to highlight the tissues surrounding the tumor better.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the feasibility of utilizing an MRI-guided tri-60Co teletherapy system for liver SBRT, as determined the treating radiation oncologist's ability to accurately visualize and align to the target lesion(s).

II. To assess the feasibility of using a three versus five fraction scheme, for one versus multiple (i.e., =< 5) target lesions.

SECONDARY OBJECTIVES:

I. To determine the tumor local control (LC), disease specific survival (DSS), and overall survival (OS).

II. To gather biomarkers that may elucidate differential immunogenic responses from the three versus the five fraction SBRT regimens.

OUTLINE:

Patients undergo MRI-guided Tri-60Co teletherapy SBRT 3-5 fractions over 1-2 weeks.

After completion of study treatment, patients are followed up at approximately 4-6 weeks, and then every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients may have either metastatic lesions from another primary site or primary hepatocellular carcinoma; patients with one histologically confirmed metastatic lesion of the liver who are presenting for local therapy for lesions concerning for metastases that cannot or should not be biopsied will also be considered for enrollment on a case by case basis; patients can simultaneously receive treatment for multiple hepatic lesions meeting the prior two requirements, at the discretion of the treating radiation oncologist
* Karnofsky performance status (KPS) >= 70
* No active infections requiring systemic antibiotics
* If a woman is of childbearing potential, a negative urine or serum pregnancy test must be documented; women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; or abstinence) for duration of study participation and for up to 4 weeks following the study
* Ability to understand and willingness to sign a written informed consent

Exclusion Criteria:

* Pregnant women, or women of childbearing potential who are sexually active and not willing/able to use medically acceptable forms of contraception for the entire study period and for up to 4 weeks after the study
* Refusal to sign the informed consent
* Patients who are participating in a concurrent treatment protocol
* Patients for whom a plan meeting institutional quality criteria cannot be designed for SBRT treatment via the MRI-guided teletherapy unit, but for whom an SBRT plan meeting institutional quality criteria can be designed for a conventional linear accelerator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-06-03 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Plan quality of the MRI guided radiotherapy vs. conventional linac radiotherapy. | Up to 2 years
  Comparing the plan quality of the MRI guided radiotherapy to conventional determined by the ability to create treatment plans that are comparable to those generated by a conventional linear accelerator, and by the treating radiation oncologist's ability to accurately visualize and align to the target lesion
Feasibility of SBRT delivery by the MRI-guided tri-60Co teletherapy system, calculated by recording the number of patients for whom plans were or were not comparable between the two modalities | Up to 2 years
Magnitude of target motion in three dimensional space as captured by real time imaging acquired by the MRI guided tri-60 Co teletherapy system | Up to 2 years
Velocity of target motion in three dimensional space as captured by real time imaging acquired by the MRI guided tri-60 Co teletherapy system | Up to 2 years
Quality of real-time image guidance provided the tri-60Co system, as defined by the treating radiation oncologist's ability to visualize the target lesion using the on-board MRI | Up to 2 tears

SECONDARY OUTCOMES:
Collection of biomarkers that may be associated with an immunologic systemic response to SBRT | Up to 2 years
DSS | Up to 2 years
Frequency of acute grade 2-5 gastrointestinal toxicity graded using the Common Toxicity Criteria version 4.0 | Up to 2 years
Infield tumor LC | Up to 2 years
OS | Up to 2 years
Validity of automatically segmented contours generated by the MRI-guided tri-60Co teletherapy system through independent evaluation of images obtained | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ann Raldow, MD, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States